CLINICAL TRIAL: NCT05074303
Title: Yeast-derived Beta-glucan Supplementation on Antibody Response Following Influenza Vaccination: A Randomized, Placebo-controlled Study (M-Unity)
Brief Title: Beta-glucan and Immune Response to Influenza Vaccine
Acronym: M-Unity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Danstar Ferment AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB202101959
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-09

CONDITIONS: Healthy Aging
Keywords: beta-glucan; influenza; immunity; antibodies
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; beta-Glucans

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Beta-glucan (Experimental): 500 mg/day beta-glucan
  Interventions: Biological: Influenza Vaccine; Dietary Supplement: Beta-glucan
- Placebo (Placebo Comparator): 500 mg/day cellulose
  Interventions: Biological: Influenza Vaccine; Dietary Supplement: Placebo

INTERVENTIONS:
Biological: Influenza Vaccine — All subjects will receive the influenza vaccine.
Dietary Supplement: Beta-glucan — 2 - 250 mg capsules/day of beta-glucan derived from Baker's yeast
  Arms: Beta-glucan
Dietary Supplement: Placebo — 2 - 250 mg capsules/day of cellulose
  Arms: Placebo

SUMMARY:
This trial in healthy adults will determine the effects of beta-glucan, a dietary fiber supplement isolated from baker's yeast, on immune response to the influenza vaccine.

DETAILED DESCRIPTION:
Beta-glucans have been shown to enhance the innate and adaptive immune responses in cell cultures, animal models, and humans, thus adults over the age of 50 years receiving the influenza vaccination may benefit in terms of their immune response from supplementation with beta-glucans. This is a 6-week randomized, double-blind, placebo-controlled, 2-arm parallel study designed to evaluate the adjuvant effect of beta-glucan dietary supplementation during influenza vaccination. Participants will consume either the beta-glucan or placebo capsules for 42 days. Participants will complete an online Qualtrics daily questionnaire of compliance, fatigue, and cold and flu symptoms throughout the 42-day study. Influenza vaccine will be administered on or about day 14. The Gastrointestinal Symptom Rating Scale (GSRS) and the Mood and Feelings Questionnaire (MFQ) will be completed at baseline, 2 weeks and 6 weeks. Blood draws for antibody and cytokine response will be completed at baseline, and on or about days 14 and 15, and on day 42.

ELIGIBILITY:
Inclusion Criteria:

1. Adult volunteers ≥ 50 years of age.
2. Planning to be vaccinated for influenza
3. Have been immunized for COVID-19
4. Willing and able to provide written informed consent in English.
5. Willing and able to comply with all the study-related procedures, including attending to study visits for blood draw, taking the influenza vaccine, intake of the study supplement, and completing study questionnaires.

Exclusion Criteria:

1. Demonstrate an inability to comply with the study-related procedures.
2. Have a history of a severe reaction or hypersensitivity following vaccination with influenza vaccine, vaccination with any other vaccine containing the same substances, or intake of the study product.
3. Have an immune system alteration because of an underlying illness (e.g., autoimmune disease) or immune-suppressing treatment (e.g., steroids (last 30 days); cytotoxic drugs, medical surgery, or radiation therapy during the 6 months, previous to enrollment).
4. Be concurrently participating in a clinical trial that, in the judgement of the investigator, would interfere with the evaluation of the study outcomes.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Food Science and Human Nutrition Department, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moreno ML, Nieves CJ, Hebert K, Vivas CA, Rivero-Mendoza D, Colee J, Tompkins TA, Dahl WJ. Yeast Beta-Glucan Enhances Antibody Response Following Influenza Vaccination - A Double-Blind, Randomized, Placebo-Controlled Pilot Trial. J Diet Suppl. 2025;22(5):795-810. doi: 10.1080/19390211.2025.2539876. Epub 2025 Jul 31. PMID 40746014

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Beta-glucan | Placebo
Started | 38 | 40
Completed | 38 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beta-glucan | Placebo | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (9) | 71 (11) | 71 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 39 | 75
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 35 | 35 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Antibody Titer
Description: Change in influenza-specific antibody influenza A titer to the influenza vaccine after beta-glucan supplementation. Titer from 0 to 1024; higher titer indicates stronger immune response.
Time Frame: 42 days (mean of Day -14 and 0 compared to Day 28)
Population: A total of 40 participants were randomized to the placebo group and 38 to the beta-glucan group over two vaccination seasons. However, the antibody titer could only be analyzed in Season 1 (19 to placebo and 24 to beta-glucan) due to an ineffective influenza antigen source, which explains the discrepancy.
Measure: Mean (Standard Deviation); unit: Titer
Arm/Group | Beta-glucan | Placebo
Number analyzed (Participants) | 24 | 19
Titer
  Baseline (Mean of Day -14 and Day 0) | 127 (105) | 143 (172)
  Intervention (Day 28) | 241 (272) | 160 (165)

2. Secondary Outcome: Inflammatory Cytokine Profile
Description: Change in IFN-γ
Time Frame: 28 days (Day 0, Day 1, and Day 28)
Population: IFN-γ was analyzed in all participants in season 1 and season 2.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Beta-glucan | Placebo
Number analyzed (Participants) | 38 | 40
pg/mL
  Day 0 | 2.3 (0.1) | 2.4 (0.4)
  Day 1 | 8.2 (1.7) | 8.3 (2.9)
  Day 28 | 3.3 (0.5) | 2.3 (0.4)

3. Secondary Outcome: Incidence of Influenza and Covid-19
Description: Self-reported incidence of influenza and Covid-19
Time Frame: 28 days
Population: This outcome was assessed on all participants in Season 1 and Season 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Beta-glucan | Placebo
Number analyzed (Participants) | 38 | 40
Participants | 0 | 0

4. Secondary Outcome: Fever
Description: Number of subjects with self-reported fever
Time Frame: 28 days
Population: This outcome was assessed on all participants in season 1 and season 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Beta-glucan | Placebo
Number analyzed (Participants) | 38 | 40
Participants | 1 | 1

5. Secondary Outcome: Cold and Flu Symptoms
Description: Score on the Modified Jackson Criteria rating scale from 0 (no symptoms) to 3 (severe symptoms).
Time Frame: 28 days
Population: Cold and flu symptoms were monitored in all participants in Seasons 1 and 2.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Beta-glucan | Placebo
Number analyzed (Participants) | 38 | 40
Score on scale | 0.92 (0.07) | 0.70 (0.06)

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Beta-glucan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT05074303/Prot_SAP_001.pdf